CLINICAL TRIAL: NCT01307280
Title: Weight Management Demonstration Project: Healthy Eating and Active Living in TRICARE Households
Brief Title: Weight Management Demonstration Project: HEALTH
Acronym: HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The Cooper Institute (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0209792; H94002-05-C-003 (Other Grant/Funding Number: Department of Defense, TRICARE Medical Activity)
Record Dates: First submitted 2011-02-22; First posted 2011-03-02 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Weight Loss
Keywords: Behavioral Weight Management Intervention; weight loss; cost-effective analysis; high blood pressure; randomized clinical trial; behavioral interventions; physical activity; dietary change; obesity
MeSH Terms: conditions — Weight Loss; Hypertension; Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Basic HEALTH (Experimental): Participants received the bookHEALTH manual and eHEALTH tools, the basic Internet component of the intervention
  Interventions: Behavioral: RCT1
- Interactive Internet (Experimental): Intervention intensity increased in RCT2, which included bookHEALTH and an interactive version of eHEALTH that provided tailored computerized feedback whenever participants submitted weekly assessments.
  Interventions: Behavioral: RCT2
- Behavioral Counseling (Experimental): RCT3 included bookHEALTH, the interactive version of eHEALTH, and telephonic coaching support provided by trained health lifestyle coaches every 2 weeks alternating between a telephone call (typically 15 to 20 minutes) and a personalized e-mail. The coaches used motivational interviewing, helped participants solve problems, and reinforced their successes.
  Interventions: Behavioral: RCT3

INTERVENTIONS:
Behavioral: RCT1 — the bookHEALTH manual and eHEALTH tools, the basic Internet component of the intervention
  Arms: Basic HEALTH
Behavioral: RCT2 — bookHEALTH and an interactive version of eHEALTH that provided tailored computerized feedback whenever participants submitted weekly assessments
  Arms: Interactive Internet
Behavioral: RCT3 — bookHEALTH, the interactive version of eHEALTH, and telephonic coaching support provided by trained health lifestyle coaches every 2 weeks alternating between a telephone call (typically 15 to 20 minutes) and a personalized e-mail. The coaches used motivational interviewing, helped participants solve problems, and reinforced their successes.
  Arms: Behavioral Counseling

SUMMARY:
The study investigated the effectiveness and cost-effectiveness of a cognitive and behavioral weight management program, complemented by an interactive Web site and brief telephone coaching, implemented among TRICARE non-active-duty beneficiaries.

A total of 1,755 participants from four Midwestern states were randomized to one of three randomized controlled trial groups with increasing intervention intensity: mailed material and basic Web access (RCT1), plus an interactive Web site (RCT2), plus brief phone- and Web-based coaching support from health lifestyle coaches (RCT3). The study assessed changes in participants' weight, blood pressure, diet, and physical activity from baseline to 6, 12, and 15 to 18 months. Analyses estimated overall cost savings and calculated the cost-effectiveness ratio of each randomized controlled trial compared with a "do-nothing" alternative as the cost per quality-adjusted life year.

DETAILED DESCRIPTION:
Lifestyle modification interventions that promote healthful eating habits and physical activity can be effective in producing weight losses of 4% to 9% of initial bodyweight. If maintained, this level of weight loss can reduce hypertension, high blood glucose, and elevated lipids. However, weight losses often plateau after 6 months, and weight regain begins after 12 months. Accordingly, there is interest in interventions, such as Web-based reinforcement and brief counseling to maintain weight loss over time and in the relative cost-effectiveness of program delivery modes.

Most obesity treatment programs focus on outcomes for individuals without assessing population-based cost savings. This study suggests that a broader perspective can help to identify the benefit of weight management in adult populations. Accordingly, this study assessed the cost-effectiveness of a weight management program in a population of adults served by a large health care system-the TRICARE Management Activity (TMA), the agency that manages the TRICARE health care benefits for active-duty service members, retired service members, their families, National Guard/Reserve members, and their families. The annual direct medical costs of overweight/obesity for beneficiaries enrolled in TRICARE Prime are estimated to exceed $1.1 billion. This study investigated the effectiveness and cost-effectiveness of methods to deliver a cognitive-behavioral weight loss intervention.

ELIGIBILITY:
Inclusion Criteria:

* TRICARE Prime non-active-duty beneficiaries
* Body Mass Index of 25 to 50
* Living in 4 midwestern states (TRICARE region)

Exclusion Criteria:

* Not able to engage in physical activity
* Pregnant
* Body mass index greater than 50
* Body mass index less than 25
* Human immunodeficiency virus infected
* current cancer

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2395 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Body Mass Index BMI | change in body mass index at baseline
BMI | change in body mass index at 6 months
BMI | change in body mass index at 12 months
BMI | change in body mass index at 18 months

SECONDARY OUTCOMES:
Blood Pressure | change in blood pressure at baseline, and 6,12,18 months

CONTACTS AND LOCATIONS:
Overall Officials: James Hersey, PhD, Principal Investigator — RTI International
Locations (3):
- United States (3):
  - RTI Study Center, Swansea, Illinois
  - RTI International, Research Triangle Park, North Carolina
  - RTI Study Center, Fairborn, Ohio

REFERENCES:
- [Derived] Hersey JC, Khavjou O, Strange LB, Atkinson RL, Blair SN, Campbell S, Hobbs CL, Kelly B, Fitzgerald TM, Kish-Doto J, Koch MA, Munoz B, Peele E, Stockdale J, Augustine C, Mitchell G, Arday D, Kugler J, Dorn P, Ellzy J, Julian R, Grissom J, Britt M. The efficacy and cost-effectiveness of a community weight management intervention: a randomized controlled trial of the health weight management demonstration. Prev Med. 2012 Jan;54(1):42-9. doi: 10.1016/j.ypmed.2011.09.018. Epub 2011 Oct 6. PMID 22001689